CLINICAL TRIAL: NCT00003875
Title: Treatment of Acute Myelogenous Leukemia With Busulfan and Etoposide Followed by Autologous or Syngeneic Stem Cell Rescue and Low-Dose Interleukin 2 (IL-2) Immunotherapy
Brief Title: Busulfan and Etoposide Followed by Peripheral Blood Stem Cell Transplant and Low-Dose Aldesleukin in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1315.00; NCI-2011-00439 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1315.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Childhood Acute Myeloid Leukemia in Remission; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Busulfan; Etoposide; aldesleukin; Interleukin-2; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemo, stem cell rescue, interleukin therapy) (Experimental): PREPARATIVE REGIMEN: Patients receive busulfan IV over 2 hours or PO every 6 hours on days -7 to -4 and etoposide IV on day -3.
  STEM CELL INFUSION: Patients undergo autologous or syngeneic PBSC rescue on day 0.
  POST-TRANSPLANT ALDESLEUKIN THERAPY: Beginning 30-100 days after transplant, patients receive low-dose aldesleukin SC daily for 12 weeks.
  Interventions: Drug: busulfan; Drug: etoposide; Biological: aldesleukin; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: busulfan — Given PO or IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Procedure: peripheral blood stem cell transplantation — Undergo autologous or syngeneic stem cell rescue
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase II trial studies the side effects and how well giving busulfan and etoposide followed by peripheral blood stem cell transplant (PBSCT) and low-dose aldesleukin works in treating patients with acute myeloid leukemia (AML). Drugs used in chemotherapy, such as busulfan and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. A PBSCT may be able to replace blood-forming cells that were destroyed by chemotherapy. This may allow more chemotherapy to be given so that more cancer cells are killed. Aldesleukin may stimulate the white blood cells to kill cancer cells. Giving busulfan and etoposide together followed by PBSCT and aldesleukin may be an effective treatment for AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity and overall survival of high dose Bu (busulfan)/VP-16 (etoposide) followed by post-transplant low-dose interleukin (IL)-2 (aldesleukin) in patients with AML.

SECONDARY OBJECTIVES:

I. To estimate the rate of relapse associated with this regimen.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive busulfan intravenously (IV) over 2 hours or orally (PO) every 6 hours on days -7 to -4 and etoposide IV on day -3.

STEM CELL INFUSION: Patients undergo autologous or syngeneic PBSC rescue on day 0.

POST-TRANSPLANT ALDESLEUKIN THERAPY: Beginning 30-100 days after transplant, patients receive low-dose aldesleukin subcutaneously (SC) daily for 12 weeks.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have AML that falls into one of the following categories:
* AML in 1st complete remission (CR) with intermediate or high risk of relapse following conventional therapy; at least, one of the following features is needed:

  * Patient required more than one cycle of induction to achieve first CR
  * White blood cell count (WBC) > 100,000/mm^3 at diagnosis
  * Any of the following cytogenetic abnormalities: inv (3), t(3:3), del (5q) or -5, 11q23, del(7q) or -7, del (20q) or -20, abnormal 12p, +11 or t8
  * Any other abnormalities or combination of abnormalities which would predict intermediate or high risk of relapse
* AML beyond first CR
* Any patient with an identical twin donor who also meets the criteria above
* Patients with AML in 1st CR should receive at least two cycles of consolidation chemotherapy prior to mobilization and transplant
* Patients must have an adequate number of stem cells previously collected (i.e., > 2 x 10^8 total nucleated cell [TNC] of bone marrow [BM]/kg or 4 x 10^6 [CD]34+ PBSC/kg, unless approved otherwise by Dr. Holmberg); prior to stem cell collection patients must be documented to be in remission and to have received two cycles of consolidation therapy after induction therapy
* Pre-Study tests have been performed
* Patient must sign an institutional review board (IRB) approved informed consent, conforming with federal and institutional guidelines

Exclusion Criteria:

* Patients with good risk AML defined by cytogenetic evaluation with these abnormalities: inversion 16 or t8;21
* Patient's life expectancy is severely limited by diseases other than AML
* Patient is human immunodeficiency virus (HIV) seropositive
* Patient is pregnant
* Patient's creatinine > 2.0 mg/dl
* Patient's total bilirubin > 2.0 mg/dl (unless Gilbert's disease)
* Or serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) >= 2.5 x upper limit of normal (ULN) not due to leukemia
* Patient has a history of congestive heart failure, uncontrolled arrhythmias or left ventricular ejection fraction (LVEF) < 50%
* Patient has an unrelated human leukocyte antigen (HLA) matched donor and is eligible for a higher priority Fred Hutchinson Cancer Research Center (FHCRC) protocol (for FHCRC patients only)
* Patient has an HLA matched or one antigen mismatch family donor available
* Patients with a significant active infection that precludes transplant
* Patients with a Karnofsky Performance Score less than 70

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-10-13 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller HN, Berger MB, Askew S, Kay MC, Hopkins CM, Iragavarapu MS, de Leon M, Freed M, Barnes CN, Yang Q, Tyson CC, Svetkey LP, Bennett GG, Steinberg DM. The Nourish Protocol: A digital health randomized controlled trial to promote the DASH eating pattern among adults with hypertension. Contemp Clin Trials. 2021 Oct;109:106539. doi: 10.1016/j.cct.2021.106539. Epub 2021 Aug 13. PMID 34400362

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy): PREPARATIVE REGIMEN: Patients receive busulfan IV over 2 hours or PO every 6 hours on days -7 to -4 and etoposide IV on day -3.
  STEM CELL INFUSION: Patients undergo autologous or syngeneic PBSC rescue on day 0.
  POST-TRANSPLANT ALDESLEUKIN THERAPY: Beginning 30-100 days after transplant, patients receive low-dose aldesleukin SC daily for 12 weeks.
  busulfan: Given PO or IV
  etoposide: Given IV
  aldesleukin: Given SC
  peripheral blood stem cell transplantation: Undergo autologous or syngeneic stem cell rescue
Period: Overall Study
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Screen Failed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 52 [26 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Patients on Busulfan and Etoposide Followed by Stem Cell Rescue and Aldesleukin
Description: Estimated by the method of Kaplan and Meier.
Time Frame: From date of transplant to date of death from any cause, assessed up to 178 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Number analyzed (Participants) | 29
Participants | 14

2. Primary Outcome: Toxicity Associated With High-dose Busulfan and Etoposide Followed by Stem Cell Rescue
Description: Toxicity is defined as any grade 3 or grade 4 toxicity per the Bearman toxicity grading criteria following Busulfan and Etoposide high-dose chemotherapy, stem cell transplant, and the inability to recover sufficiently by day 100 to start IL-2 therapy.
Time Frame: Day -7 of transplant to 100 days post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Number analyzed (Participants) | 29
Participants | 2

3. Primary Outcome: Toxicity Associated With Aldesleukin Treatment After Stem Cell Rescue
Description: Toxicity during IL-2 therapy of any of the following per NCI Common Toxicity version 3: grade 2, 3, 4, or 5 CNS (except grade 0-3 malaise, fatigue, anxiety and depression) toxicity; grade 3, 4, or 5 non-CNS or non-hematologic toxicity; any grade 4 or 5 hematologic toxicity.
Time Frame: IL-2 administration to one month after completion of IL-2 treatment
Population: 29 patients underwent autologous transplant and 21 of these patients after transplant went on to get IL-2 treatment . Toxicity for IL-2 therapy thus was only analyzed in these later 21 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Number analyzed (Participants) | 21
Participants | 6

4. Secondary Outcome: Proportion of Patients Who Relapsed Associated With the Regimen
Time Frame: From date of transplant to date of death from any cause, assessed up to 178 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Stem Cell Rescue, Interleukin Therapy)
Number analyzed (Participants) | 29
Participants | 16

ADVERSE EVENTS:
Time Frame: Day -7 pre transplant to approximately 212 days post transplant
Description: Transplant (TX) toxicities grade ≥3 per Bearman toxicity grading measured day -7 to the start of IL-2 therapy.
  Post-TX IL-2 therapy toxicities graded per NCI Common Toxicity version 3 measured from the start of IL-2 to one month after completion of IL-2: grade 2-5 CNS (except grade 0-3 malaise, fatigue, anxiety and depression) toxicity; grade 3- 5 non-CNS or non-hematologic toxicity; any grade 4 or 5 hematologic toxicity. 29 patients got TX and 21 patients got IL-2 after transplant.
Groups:
- Treatment: PREPARATIVE REGIMEN: Patients receive busulfan IV over 2 hours or PO every 6 hours on days -7 to -4 and etoposide IV on day -3.
  STEM CELL INFUSION: Patients undergo autologous or syngeneic PBSC rescue on day 0.
  POST-TRANSPLANT ALDESLEUKIN THERAPY: Beginning 30-100 days after transplant, patients receive low-dose aldesleukin SC daily for 12 weeks.
  busulfan: Given PO or IV
  etoposide: Given IV
  aldesleukin: Given SC
  peripheral blood stem cell transplantation: Undergo autologous or syngeneic stem cell rescue
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 5/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=29)
Hospitalization for pulmonary embolus (likely from Hickman line) (Vascular disorders) | 1 — Transplant toxicity. Note: No SAEs in IL-2 portion of the study.
Prolonged Hospitalization (34 days) for hyperbilirubinemia (Investigations) | 1 — Transplant toxicity. Note: No SAEs in IL-2 portion of the study. Possible autoimmune hemolysis or syngeneic GVHD and severe skin desquamation
Hospitalization for infection (Infections and infestations) | 2 — Transplant toxicity. Note: No SAEs in IL-2 portion of the study.
Stroke (Nervous system disorders) | 1 — Transplant toxicity. Note: No SAEs in IL-2 portion of the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment (N=29)
Myelosuppression (Blood and lymphatic system disorders) | 29 — Transplant toxicity
Hematologic (Blood and lymphatic system disorders) | 4/21 — NCI Common Toxicity Version 3 - Toxicity to IL-2 Therapy. Only 21 of 29 transplanted patients got IL-2 therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No